CLINICAL TRIAL: NCT07223593
Title: A Study to Investigate the Efficacy and Safety of Orforglipron Once Daily in Participants With Peripheral Artery Disease: A Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Efficacy and Safety of Orforglipron in Participants With Peripheral Artery Disease
Acronym: ATTAIN-PAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27632; 2025-523283-21-00 (EU CTIS Number); J2A-MC-GZPR (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect and safety of orforglipron once daily in participants with Fontaine II peripheral arterial disease (PAD). Participation in the study will last about 58 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have symptomatic PAD with intermittent claudication of Fontaine Stage II
* Have an Ankle Brachial Index (ABI) of 0.9 or less

Exclusion Criteria:

* Have a body mass index (BMI) less than 23 kilogram per square meter (kg/m2)
* Have Hemoglobin A1c (HbA1c) greater than 10%
* Have walking ability limited by conditions other than PAD
* Have a planned lower limb surgery or any other surgery affecting walking ability
* Had peripheral revascularization procedure within 90 days prior to the day of screening or planning to undergo peripheral revascularization during the clinical trial
* Had stroke, transient ischemic attack, myocardial infarction, coronary or carotid revascularization, or hospitalization for unstable angina pectoris within 60 days prior to screening
* Have heart failure presently classified as being in New York Heart Association class III - IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Maximum Walking Distance | Baseline, Week 52
  On a constant load treadmill test

SECONDARY OUTCOMES:
Percent Change from Baseline in Pain Free Walking Distance | Baseline, Week 52
  On a constant load treadmill test
Change from Baseline in Vascular Quality of Life (VascuQoL-6) Questionnaire Score | Baseline, Week 52
Change from Baseline in 6 Minute Walk Test Distance (meters) | Baseline, Week 52
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 52
Change from Baseline in Systolic Blood Pressure (mmHg) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (138):
- United States (30):
  - St. Vincent's Birmingham Hospital, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Axsendo Clinical Research - Peak Heart & Vascular - Surprise, Surprise, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Valley Clinical Trials, Inc., Northridge, California
  - The Cardiovascular Center, Redding, California
  - InvivoCure, Van Nuys, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Lakeview Institute of Clinical Research, Leesburg, Florida
  - Inpatient Research Clinic, Miami Lakes, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - St Johns Center for Clinical Research, Saint Augustine, Florida
  - ASHA Clinical Research - Munster, LLC, Hammond, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Deaconess Clinic- Gateway, Newburgh, Indiana
  - Flourish Research - Bowie, Bowie, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - The Jackson Clinic, Jackson, Tennessee
  - East Coast Institute for Research - Jefferson City, Jefferson City, Tennessee
  - Biopharma Informatic, LLC, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Sherman Clinical Research, Sherman, Texas
  - NextStage Clinical Research - Waco, Waco, Texas
  - Alpine Research Organization, Clinton, Utah
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia
  - ERA Health Research - CardioNow - Lynnwood, Lynnwood, Washington
  - Eastside Research Associates, Redmond, Washington
- Argentina (9):
  - CIPREC, Buenos Aires
  - Sanatorio Finochietto, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - DIM Clínica Privada, Ramos Mejía
  - INECO Neurociencias Oroño, Rosario
  - Instituto de Investigaciones Clinicas Rosario, Rosario
  - Go Centro Medico San Nicolás, San Nicolás
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
- Australia (6):
  - Box Hill Hospital, Box Hill
  - Core Research Group, Brisbane
  - Canberra Hospital, Canberra
  - University of the Sunshine Coast (UniSC) Clinical Trials - Meadowbrook, Meadowbrook
  - Royal Perth Hospital, Perth
  - Gold Coast University Hospital, Southport
- Brazil (8):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Hospital Universitário João de Barros Barreto, Belém
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Universidade Federal de Goias, Goiânia
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Centro Avançado De Pesquisa, Estudos E Diagnóstico (CAPED) - Centro Médico RibeirãoShopping, Ribeirão Preto
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí
- Canada (7):
  - THEO Medical Concorde, Laval
  - Alpha Recherche Clinique - Lévis, Lévis
  - KMH Cardiology Centres - Stoney Creek, Stoney Creek
  - Corcare, Toronto
  - Unity Health Toronto, St. Michael's Hospital, Toronto
  - Toronto General Hospital, Toronto
  - Cardio 1 Medical Clinic, Winnipeg
- China (15):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Heilongjiang Provincial Hospital, Harbin
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Nanjing First Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital,Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin People' s Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an
- France (7):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - CHRU Troussau, Chambray-lès-Tours
  - Hôpital Saint Philibert, Lomme
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Groupe hospitalier Paris saint Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
- India (8):
  - Jawaharlal Nehru Medical College, Aligarh
  - M. P. Birla Group - Belle Vue Clinic, Kolkata
  - Government Medical College - Kozhikode, Kozhikode
  - Lata Mangeshkar Hospital - Digdoh, Nagpur
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - Vijan Hospital & Research Centre, Nashik
  - Sir Ganga Ram Hospital, New Delhi
  - All India Institute of Medical Sciences - Rishikesh, Rishikesh
- Japan (23):
  - University of Yamanashi Hospital, Chūō
  - Fukuyama City Hospital, Fukuyama
  - Hakodate Municipal Hospital, Hakodate
  - Medical Corporation Sapporo Heart Center Sapporo Cardio Vascular Clinic, Higashi
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Shinyurigaoka General Hospital, Kawasaki
  - Kokura Memorial Hospital, Kitakyushu
  - Kobe City Medical Center General Hospital, Kobe
  - Seikeikai Medical Corporation New Tokyo Heart Clinic, Matsudo
  - Tokyo Saiseikai Central Hospital, Minatoku
  - Japanese Red Cross Musashino Hospital, Musashino-shi
  - Koujunkai Daido Clinic, Nagoya
  - Nakakinen clinic, Naka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Keisatsu Hospital, Osaka
  - Kansai Electric Power Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Saitama City Hospital, Saitama
  - Japan Community Healthcare Organization Hokkaido Hospital, Sapporo
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho
  - Municipal Toyonaka Hospital, Toyonaka
  - Yamagata University Hospital, Yamagata
  - Yokohama City Minato Red Cross Hospital, Yokohama
- Netherlands (3):
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Radboudumc, Nijmegen
- Poland (5):
  - Centrum Medyczne INTERCOR Sp. z o.o., Bydgoszcz
  - NZOZ Twoje Zdrowie EL Sp. z o. o., Elblag
  - Przychodnie Grudziądz, Grudziądz
  - Centrum Medyczne Komorniki, Komorniki
  - Poliklinika Kardiologiczna Serce, Leszno
- Research and Cardiovascular Corp., Ponce, Puerto Rico
- Slovakia (2):
  - Alian - Bardejov, Bardejov
  - MEDIVASA, Žilina
- South Korea (4):
  - Daegu Catholic University Medical Center, Daegu
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (6):
  - Leeds General Infirmary, Leeds
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London
  - Derriford Hospital, Plymouth
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Swansea University, Swansea
  - Moorgreen Hospital, West End

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Efficacy and Safety of Orforglipron in Participants With Peripheral Artery Disease (ATTAIN-PAD) — https://trials.lilly.com/en-US/trial/663317